## Plication of Fascia Transversalis and Its Role in Reduction of Seroma Formation Post Laparoscopic Transabdominal Preperitoneal Repair of Direct Inguinal Hernia

A Thesis Submitted For Partial Fulfillment of MSc Degree of General Surgery

Ву

Dr. Mohammed Elshwadfy Nageeb Abdelaziz

Ethical Approval Number: MS 204-2024

## Supervisors

Prof. Dr. George Abdelfady Nashed Professor of General Surgery Faculty of Medicine, Cairo University

Dr. Khaled Mosleh Mohammed Torfa Lecturer of General Surgery Faculty of Medicine, Cairo University

Dr. Mohammed Elshwadfy Nageeb Abdelaziz Lecturer of General Surgery Faculty of Medicine, Cairo University

> Faculty of Medicine Cairo University 2025

## Statistical Analysis

Data are analyzed using SPSS version 21. Descriptive statistics are presented as means with standard deviation for continuous variables and frequencies with percentages for categorical variables. Comparisons between groups are made using:

- Chi-square test or Fisher 's exact test for categorical data.
- Student 's t-test for normally distributed continuous variables.
- Mann-Whitney U test for non-normally distributed data.
- Paired t-test for preoperative and postoperative comparisons within each group.
- Pearson or Spearman correlation tests to assess relationships between variables.

A p-value 0.05 is considered statistically significant.

## **Ethical Considerations**

This study is conducted in accordance with the Declaration of Helsinki and is approved by the Institutional Review Board (IRB) of Cairo University. Written informed consent is obtained from all participants prior to enrollment. Patients' confidentiality is maintained, and their data are anonymized. No financial incentives are provided, and participation is voluntary. Potential risks, including coagulation alterations and allergic reactions, are clearly explained to the patients.